CLINICAL TRIAL: NCT01629472
Title: Protection From Gender-based Violence in Cote d'Ivoire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Innovations for Poverty Action (Other); International Rescue Committee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1007007040
Record Dates: First submitted 2012-06-13; First posted 2012-06-27 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Domestic Violence; Family and Household
Keywords: Gender norms; Financial Autonomy; Economic Well-being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSLA + gender dialogue groups: treatment (Experimental)
  Interventions: Behavioral: VSLA + Gender dialogue groups
- VSLA only: control (Active Comparator)
  Interventions: Behavioral: VSLA + Gender dialogue groups

INTERVENTIONS:
Behavioral: VSLA + Gender dialogue groups — Dialogue groups discussing household discussion making and gender norms facilitated by IRC.

SUMMARY:
There is some evidence that suggests that economic empowerment and challenging gender inequalities and prevailing ideas on masculinities will lead to a decrease in levels of partner violence. However, there is still a gap in our understanding of what elements are required. This project evaluates whether participation within a savings group and a discussion group confronting gender norms will lead to an increase in women's individual agency and decision-making ability that will improve their economic independence and decrease intimate partner violence in their homes.

ELIGIBILITY:
Inclusion Criteria:

* No Prior experiences with microcredit programs
* 18+
* Source of stable income

Exclusion Criteria:

* 18+
* prior experience with microcredit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 981 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess differences in past year, self-reported intimate partner violence (physical and sexual)between treatment and control groups. This will be assessed using the CTS-2 scale | 24 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: jhumka gupta, ScD, Principal Investigator — Yale University
Locations (1):
- International Rescue Committee, Abidjan, Côte d’Ivoire

REFERENCES:
- [Result] Gupta J, Falb K, Kpebo D, Annan J. Abuse from in-laws and associations with attempts to control reproductive decisions among rural women in Cote d'Ivoire: a cross-sectional study. BJOG. 2012 Aug;119(9):1058-66. doi: 10.1111/j.1471-0528.2012.03401.x. Epub 2012 Jun 7. PMID 22676807
- [Derived] Blay-Tofey M, Lee BX. Preventing gender-based violence engendered by conflict: The case of Cote d'Ivoire. Soc Sci Med. 2015 Dec;146:341-7. doi: 10.1016/j.socscimed.2015.10.009. Epub 2015 Oct 14. PMID 26482357
- [Derived] Gupta J, Falb KL, Lehmann H, Kpebo D, Xuan Z, Hossain M, Zimmerman C, Watts C, Annan J. Gender norms and economic empowerment intervention to reduce intimate partner violence against women in rural Cote d'Ivoire: a randomized controlled pilot study. BMC Int Health Hum Rights. 2013 Nov 1;13:46. doi: 10.1186/1472-698X-13-46. PMID 24176132